CLINICAL TRIAL: NCT05356377
Title: A Preliminary Study of the Neurological and Neuropsychological Effects of Palynziq-Related Changes in Phenylalanine in Individuals With Phenylketonuria (PKU)
Brief Title: Preliminary Study of Brain Effects of Palynziq-Related Changes in Phenylalanine in Individuals With PKU
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Shawn Christ, Associate Professor, University of Missouri-Columbia
Other Study IDs: 2055562
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PKU Palynziq Group: Individuals with PKU who have previously completed baseline (pre-Palnyziq) neurocognitive and neuroimaging evaluations and have since demonstrated a significant and prolonged Phe response to Palynziq (as reflected by at least 3 consecutive months of Phe levels below 360 μmol/L).
  Interventions: Drug: Pegvaliase-Pqpz

INTERVENTIONS:
Drug: Pegvaliase-Pqpz — Participants will have been prescribed pegvaliase-pqpz (Palynziq) by their primary metabolic care providers as part of their standard care. [Note that prescription and standard care are independent of the present study.]

SUMMARY:
The goal of the proposed study is to elucidate neurologic and neuropsychological improvements associated with Palynziq-related reduction in plasma Phe levels in individuals with PKU. To this end, investigators will utilize state-of-the-art neuropsychological and multi-modal neuroimaging methods to examine the effects of large Phe level reduction (levels <360 μmol/L for at least 3 consecutive months) on GM and WM brain structures, brain concentrations of Phe, functionality of brain networks, and associated cognitive functioning in a sample of individuals with PKU who are being treated with Palyzniq.

DETAILED DESCRIPTION:
Past studies have documented PKU-related disruptions in brain phenylalanine (Phe) levels, white matter (WM) and gray matter (GM) brain structures, functional connectivity, and neurocognitive functioning. Additional research suggests that the disruptive effects of excessive blood Phe levels likely contribute to these abnormalities, and treatment aimed at lower Phe levels may lead to significant improvements.

Within this context, the primary aim is to test the hypotheses that Palynziq-related reductions in blood Phe levels will be associated with:

1. A decrease in brain Phe levels as measured by magnetic resonance spectroscopy (MRS).
2. A decrease in the extent and severity of WM abnormalities as evidenced by increased mean diffusivity values - a measure of microstructural WM integrity that is derived via diffusion-weighted magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI).
3. Closer-to-normal volumetric measurements for GM structures. Nature of this effect will be dependent on structure. For example, PKU is associated with increased volume in basal ganglia but decreased volume in posterior cortex and cerebellum (Aldridge et al., 2020; Bodner et al., 2012; Christ et al., 2016).
4. An increase in functional connectivity within the brain's functional networks as measured by resting state functional MRI (fMRI).
5. Improved performance on neurocognitive tests of executive function, attention, processing speed, and motor control.

To accomplish this aim, a total sample of up to 13 adults with PKU who have previously completed baseline (pre-Palnyziq) neurocognitive and neuroimaging evaluations will be recruited from the two sites (University of Missouri, Boston Children's Hospital). Participants will be reassessed following a significant and prolonged Phe response to Palynziq (as reflected by at least 3 consecutive months of Phe levels below 360 μmol/L).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Participants identified by newborn screening with PKU as evidenced by a blood Phe level ≥ 360μmol/L; received treatment within the first 30 days of life
* Previously received a neuropsychological and neuroimaging evaluation (as part of previously described MU or BCH studies) prior to enrollment in the present study (while Palynziq-naïve).
* Capable of providing informed consent
* Presently being treated with Palynziq and has demonstrated a prolonged Phe response to Palynziq (as reflected by at least 3 consecutive months of Phe levels below 360 μmol/L)

Exclusion Criteria:

* History of major neurologic disorder unrelated to PKU
* Contraindications for safe MRI participation such as (a) pregnancy or plans to become pregnant during period of study enrollment; or (b) metallic objects inside the body (e.g., surgical staples left in the body following surgery, middle ear prosthesis, metal foreign objects lodged inside the eye, heart pacemakers).
* Current participation in an interventional clinical trial (not Palynziq-related).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants who meet 3 primary criteria: (1) have previously completed baseline (pre-Palynziq) neurocognitive & neuroimaging evaluations as part of other studies at University of Missouri of Boston Children's Hospital, (2) have since been prescribed Palnyziq by their primary metabolic care providers, and (3) have demonstrated a prolonged blood phe response to Palynziq as reflected by 3+ months of phe levels below 360 umol/L.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Neurologic Integrity | Single timepoint for 1 hour
  Brain phenylalanine (Phe) levels, white matter integrity, gray matter integrity, functional connectivity as measured using magnetic resonance imaging (MRI)
Neuropsychological Functioning | Single timepoint for 2 hours
  Neuropsychological functioning as assessed using a comprehensive battery of standardized neuropsychological tests

SECONDARY OUTCOMES:
Cookie Theft Picture Test | Single timepoint for 10 minutes
  Verbal linguistics as assessed using the Cookie Theft Picture Test from the Boston Diagnostic Aphasia Exam
In-the-moment Psychoemotional Symptomatology | 30 minutes total per day for 7 consecutive days
  Cell phone-based ecological momentary assessment (EMA) to measure in-the-moment psychoemotional symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Christ, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: Undecided